CLINICAL TRIAL: NCT00869063
Title: A Randomized, Double-Blind, Placebo-Controlled Study of the Efficacy and Safety of a Diclofenac Sodium Patch for the Topical Treatment of Acute Pain Due to Mild to Moderate Wrist Sprain, Strain or Contusion
Brief Title: Diclofenac Patch for the Treatment of Acute Pain Due to Mild to Moderate Wrist Sprain, Strain or Contusion
Acronym: WIND
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cerimon Pharmaceuticals (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Shaily J. Reichert, V.P. of Clinical Development, Cerimon Pharmaceuticals, inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DCF-005
Record Dates: First submitted 2009-03-24; First posted 2009-03-25 (Estimated); Last update posted 2010-01-28 (Estimated); Status verified 2010-01

CONDITIONS: Acute Pain
Keywords: wrist; sprain; strain; contusion; diclofenac; patch; acute pain; acute pain due to mild to moderate wrist sprain, strain or contusion
MeSH Terms: conditions — Acute Pain; Sprains and Strains; Contusions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diclofenac Sodium Patch (Experimental)
  Interventions: Drug: Diclofenac Sodium Patch
- Placebo Patch (Placebo Comparator)
  Interventions: Drug: Matching Placebo Patch

INTERVENTIONS:
Drug: Diclofenac Sodium Patch — Topical 1% diclofenac sodium patch, applied once daily for 7 days
  Arms: Diclofenac Sodium Patch
Drug: Matching Placebo Patch — Matching placebo patch, containing identical constituents to the active drug arm except for diclofenac sodium; applied once daily for 7 days
  Arms: Placebo Patch

SUMMARY:
The purpose of the study is to assess the effectiveness of once daily application of a diclofenac sodium topical patch in reducing acute pain due to mild to moderate wrist sprain, strain or contusion when applied to the painful area.

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled, parallel group study will be conducted in patients with a mild to moderate wrist sprain, strain or contusion.

Eligible patients will be randomized (in a 1:1 ratio) to receive double-blind treatment to either the diclofenac topical patch or a matching placebo patch to be applied once daily for 7 days. Patients will return to the clinic for assessments on Day 3 and Day 7; a follow-up assessment will be conducted on Day 14. Patients will complete an electronic diary in which assessments including pain intensity, pain relief and functional disability will be recorded twice daily. Ratings of the quality of sleep will also be recorded in the diary each morning, and the use of study treatment and rescue medication will be recorded in the diary each day.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects 17 - 75 years of age
* Sustained recent, painful unilateral mild to moderate wrist sprain, strain or contusion
* Meet baseline pain criterion

Exclusion Criteria:

* Open wound or infection at the site of injury
* Severe wrist injury or wrist fracture
* Presence or history of hand, wrist or forearm nerve impingement or palsies
* Use of NSAIDs or opioids within 12 - 24 hours of wrist injury
* Presence or history of peptic ulcers or GI bleeding
* History of intolerance to NSAIDs, acetaminophen, adhesives
* Positive pregnancy test
* Positive drug screen

Ages: 17 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2009-02; Primary Completion 2009-07 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Change in average pain during daily activity | Day 3

SECONDARY OUTCOMES:
Change in average pain during daily activity | Day 7

CONTACTS AND LOCATIONS:
Locations (1):
- PPD, Austin, Texas, United States